CLINICAL TRIAL: NCT01139073
Title: A New Portable Monitor for Measuring Odorous Compounds in Oral, Exhaled and Nasal Air
Status: Completed | Type: Observational
Sponsor: Okayama University (Other)
Other Study IDs: MMorita-BB
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Halitosis
Keywords: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The B/B Checker, a new portable device for detecting odorous compounds in oral, exhaled, and nasal air, is now available. As a single unit, this device is capable of assessing several kinds of gases mixed with volatile sulfur compounds (VSCs) in addition to other odorous gasses. The purpose of the present study was to evaluate the effectiveness of the B/B Checker for detecting the malodor level of oral, exhaled, and nasal air.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oral malodor

Exclusion Criteria:

* Smoker
* Medical disorders
* Undergoing any antibiotic or other antimicrobial therapy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were recruited at the Clinic of Preventive Dentistry, Okayama University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-05; Study Completion 2010-04 (Actual)

REFERENCES:
- [Derived] Tamaki N, Kasuyama K, Esaki M, Toshikawa T, Honda S, Ekuni D, Tomofuji T, Morita M. A new portable monitor for measuring odorous compounds in oral, exhaled and nasal air. BMC Oral Health. 2011 Apr 20;11:15. doi: 10.1186/1472-6831-11-15. PMID 21504624